CLINICAL TRIAL: NCT05688033
Title: Dosimetric Limitation of Pelvic Bone and Peritoneal Space in Rectal Cancer Patients During During Neoadjuvant Chemoradiation With Capecitabine and Irinotecan
Brief Title: Dosimetric Limitation of Pelvic Bone and Peritoneal Space in Rectal Cancer Patients During Chemoradiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMRTGI0001
Record Dates: First submitted 2020-10-29; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): peritoneal space V15<850cc，pelvic bone V10<80% and normal dosimetric limitation
  Interventions: Radiation: dosimetric limitation of pelvic bone and peritoneal space during radiotherapy
- control arm (No Intervention): normal dosimetric limitation

INTERVENTIONS:
Radiation: dosimetric limitation of pelvic bone and peritoneal space during radiotherapy — dosimetric limitation of pelvic bone and peritoneal space during radiotherapy
  Arms: experimental arm

SUMMARY:
This project first retrospectively analyzes the intestinal dose indicators related to the concurrent radiotherapy and chemotherapy of rectal cancer and gastrointestinal toxicity, and the pelvic dose indicators related to hematological toxicity, and then prospectively conducts radiotherapy based on the dose indicators most closely related to toxicity. The dose is limited when the plan is made to reduce the gastrointestinal and hematological toxicity of rectal cancer with concurrent radiotherapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with rectal adenocarcinoma
2. Clinical staged T3/4 or any node-positive disease
3. Age of 18-75 years
4. Karnofsky Performance Status > 80
5. Adequate bone marrow reserve, renal and hepatic functions
6. Without previous antitumoural chemotherapy
7. No evidence of metastatic disease
8. Written informed consent before randomization
9. UGT1A1's genotype of 6/6 or 6/7

Exclusion Criteria:

1. Clinical staged I or IV
2. Age of <18 or >75 years
3. Karnofsky Performance Status < 80
4. Previous pelvis radiotherapy
5. Previous antitumoural chemotherapy
6. Clinically significant internal disease
7. Refuse to write informed consent before randomization
8. UGT1A1's genotype of 7/7

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | up to 3 years

SECONDARY OUTCOMES:
Number of Participants in Who Experienced Tumor Down-staging | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No